CLINICAL TRIAL: NCT00005828
Title: A Phase II Trial of Green Tea Extract in the Treatment of Androgen-Independent Metastatic Prostate Cancer
Brief Title: Green Tea Extract in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9951; CDR0000067842 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-06-02; First posted 2004-04-20 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- green tea extract (Experimental): Patients receive oral green tea extract six times daily for 4 months. Patients with a 50% decline in PSA, complete or partial response, or stable disease after 4 months continue treatment in the absence of disease progression or unacceptable toxicity. Patients with disease progression after 4 months receive no further treatment. Patients are followed every 3 months for 5 years or until disease progression. If disease progression, patients are followed every 6 months for 5 years.
  Interventions: Dietary Supplement: green tea extract

INTERVENTIONS:
Dietary Supplement: green tea extract

SUMMARY:
RATIONALE: Green tea extract contains substances that may slow the growth of certain cancers and may prevent the development of new cancers.

PURPOSE: Phase II trial to determine the effectiveness of green tea extract in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effectiveness and toxicity of green tea extract in patients with androgen-independent metastatic prostate cancer. II. Determine the response rate and response duration in patients treated with this regimen. III. Determine whether a decline in prostate-specific antigen (PSA) coincides with evidence of disease regression in these patients.

OUTLINE: Patients receive oral green tea extract six times daily for 4 months. Patients with a 50% decline in PSA, complete or partial response, or stable disease after 4 months continue treatment in the absence of disease progression or unacceptable toxicity. Patients with disease progression after 4 months receive no further treatment. Patients are followed every 3 months for 5 years or until disease progression. If disease progression, patients are followed every 6 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Clinically proven androgen-independent metastatic prostate cancer Radiological, physically palpable, and/or biochemical evidence of progression Increase in PSA after orchiectomy or hormonal treatment No symptoms directly attributable to metastatic disease No CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2 times upper limit of normal Cardiovascular: No uncontrolled high blood pressure No unstable angina No symptomatic congestive heart failure No uncontrolled cardiac arrhythmias No myocardial infarction in past 6 months Other: No other malignancy within the past 5 years except basal cell skin cancer No uncontrolled diabetes mellitus or inability to tolerate high sugar content of green tea at discretion of oncologist No other medical or psychiatric conditions that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior flutamide or megestrol At least 6 weeks since prior longer-acting hormonal agents such as bicalutamide At least 4 weeks since prior hormonal therapy, except luteinizing hormone- releasing hormone agonist No concurrent hormonal therapy, including corticosteroids for cancer treatment Radiotherapy: No concurrent radiotherapy Surgery: See Disease Characteristics Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2000-12; Primary Completion 2003-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Response rate and duration | Up to 5 years
Disease-regression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (16):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Jatoi A, Ellison N, Burch PA, Sloan JA, Dakhil SR, Novotny P, Tan W, Fitch TR, Rowland KM, Young CY, Flynn PJ. A phase II trial of green tea in the treatment of patients with androgen independent metastatic prostate carcinoma. Cancer. 2003 Mar 15;97(6):1442-6. doi: 10.1002/cncr.11200. PMID 12627508